CLINICAL TRIAL: NCT04836455
Title: Impact of The Real Cost Vaping Prevention Advertisements on Adolescents
Brief Title: Impact of Vaping Prevention Advertisements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-3174; 1R01CA246600-01 (NIH)
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Real Cost vaping prevention ads - Health effects theme (Experimental)
  Interventions: Behavioral: The FDA's The REal Cost vaping prevention ads - Health harms theme
- The Real Cost vaping prevention ads - Addiction theme (Experimental)
  Interventions: Behavioral: The FDA's The Real Cost vaping prevention ads - Addiction theme
- Neutral vaping ads (Other)
  Interventions: Behavioral: Neutral vaping ads

INTERVENTIONS:
Behavioral: The FDA's The REal Cost vaping prevention ads - Health harms theme — Three vaping prevention video ads from the FDA's The Real Cost prevention campaign about the health harms of vaping will be shown to participants at weeks 0, 1, and 2. Ads will be shown in a random order.
  Arms: The Real Cost vaping prevention ads - Health effects theme
Behavioral: The FDA's The Real Cost vaping prevention ads - Addiction theme — Three vaping prevention video ads from the FDA's The Real Cost prevention campaign about vaping addiction will be shown to participants at week 0, 1, and 2. Ads will be shown in a random order.
  Arms: The Real Cost vaping prevention ads - Addiction theme
Behavioral: Neutral vaping ads — Three neutral (i.e., purely informational and without graphics) vaping video ads developed by the Investigators will be shown to participants at weeks 0, 1, and 2. Ads will be shown in a random order.
  Arms: Neutral vaping ads

SUMMARY:
The purpose of this randomized controlled trial is to determine whether exposure to vaping prevention advertisements (ads) reduce susceptibility to vaping among adolescents. Previous studies have been informative, but they have tended to be one-time experimental studies that do not replicate the repeated exposures to ads that people have in the real world. This study addresses this issue by repeatedly exposing participants to vaping prevention ads over time. Participants will be adolescents aged 13-17 who currently vape or who are susceptible to vaping.

Participants will be randomly assigned to ad stimuli. They will be assigned to one of two The Real Cost trial arms-health harms or addiction-or to a control trial arm (probability of assignment is 1/3 for all trial arms). Participants in the study will take 4 online surveys over a 3-week period, once per week (At week 0, 1, 2, and 3). All participants will view randomized ad stimuli based on their trial arm and answer surveys items at each session.

DETAILED DESCRIPTION:
Tobacco prevention mass media campaigns are a key tool for reducing tobacco use among adolescents. While vaping has increased greatly among adolescents, there has been a dearth of research on effective communication strategies to reduce vaping. This study will test the impact of advertisements from the Food and Drug Administration's The Real Cost campaign on reducing susceptibility to vaping in a randomized controlled trial, illuminating whether such ads are effective as well as what themes are most effective (i.e., health harms, addiction). The investigators focus on adolescents (ages 13-17) who currently vape or are at risk of vaping.

Setting: The trial will be a longitudinal online study with 4 surveys over a 3 week period - 1 survey per week.

Recruitment: Adolescent participants will be recruited through Qualtrics, an online survey panel platform. Interested prospective participants will complete a screening questionnaire to determine their eligibility. If eligible, Qualtrics will invite them to enroll in the trial.

Informed Consent: Qualtrics will obtain parental consent online for adolescents who are eligible and interested in participating. After parental consent, adolescents will provide online assent prior to taking the survey.

Randomization: After providing informed assent, Qualtrics survey software will randomly assign participants to one of the three trial arms. Participants will have an equal chance of being randomized to any of the 3 trial arms.

Assessment: Participants in the study will take 4 surveys over a 3-week period. This will allow for multiple exposures to campaign ads. At week 0, randomize participants will be randomized to 1 of 2 FDA The Real Cost vaping prevention ad trial arms (health harms or addiction) or to a control arm (investigator created neutral ads about vaping). In each condition, participants will view 3 ads at each session, in a random order, corresponding to the theme they were assigned. At the first session (week 0), each participant will complete measures of vaping and smoking behavior, and will then view the ads that correspond to their trial arm. They will complete measures assessing message reactions after viewing each ad, followed by measures of susceptibility to vaping, vaping and smoking beliefs, and finally questions assessing demographics. For week 1 and 2 assessments, participants will complete measures of susceptibility to vaping, vaping and smoking beliefs, and vaping and smoking behavior. They will then view the same 3 ads from their trial arm and complete the message reactions measures. For the week 3 assessment, participants will only complete measures of susceptibility to vaping, vaping and smoking beliefs, and vaping and smoking behavior. Each survey will take approximately 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 13-17 years old
* Be able to read and speak English
* Be able to take an online survey in English
* Be susceptible to vaping

Exclusion Criteria:

* None

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1565 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Noar, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Kieu T, Ma H, Rohde JA, Gottfredson O'Shea N, Hall MG, Brewer NT, Noar SM. Understanding Potential Mechanisms of Vaping Prevention Messages: A Mediation Analysis of the Real Cost Campaign Advertisements. Health Educ Behav. 2025 Feb;52(1):102-112. doi: 10.1177/10901981241278565. Epub 2024 Sep 29. PMID 39342464
- [Derived] Noar SM, Gottfredson NC, Kieu T, Rohde JA, Hall MG, Ma H, Fendinger NJ, Brewer NT. Impact of Vaping Prevention Advertisements on US Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2236370. doi: 10.1001/jamanetworkopen.2022.36370. PMID 36227597

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Trial Group: This group consists of participants who took part in the pilot phase of the trial prior to its full launch. The purpose of this phase was to pilot test the clinical trial processes and procedures. Participants were recruited separately and not a part of the actual clinical trial.
Period: Overall Study
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads | Pilot Trial Group
Started | 504 | 506 | 504 | 51
Completed | 445 | 451 | 450 | 51
Not Completed | 59 | 55 | 54 | 0

BASELINE CHARACTERISTICS:
Population: The pilot trial group consists of participants who participated in the pilot phase of the trial before its full launch. The purpose of this phase was to assess how the actual clinical trial operates. Therefore, participants were recruited separately and were not part of the actual randomized clinical trial. Consequently, their outcomes are not our primary interest, and their data are not included in the final analyses reported here (e.g., total mean susceptibility to vaping).
Groups:
- Total: Total of all reporting groups
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads | Pilot Trial Group | Total
Number analyzed (Participants) | 504 | 506 | 504 | 51 | 1565
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.21 (1.17) | 15.18 (1.19) | 15.28 (1.18) | 15.55 (1.30) | 15.22 (1.18)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The following data do not include participants who identified themselves as a gender identity other than male or female.
  Participants
    number analyzed (Participants) | 498 | 497 | 503 | 51 | 1549
    Female | 126 | 122 | 110 | 22 | 380
    Male | 372 | 375 | 393 | 29 | 1169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 5 | 3 | 6 | 0 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 0 | 0 | 4
  Black or African American | 137 | 116 | 118 | 13 | 384
  White | 345 | 367 | 369 | 38 | 1119
  More than one race | 12 | 13 | 8 | 0 | 33
  Unknown or Not Reported | 2 | 5 | 3 | 0 | 10
Susceptibility to vaping [Mean (Standard Deviation); unit: units on a scale] — The 3-item Susceptibility to Vaping Scale assesses the extent to which adolescents are open to vaping, using a 1 to 4 response option scale. Here, 1 indicates the lowest susceptibility to vaping, and 4 represents the highest, with higher values indicating a greater susceptibility to vaping - essentially, a worse outcome. The overall scale score is determined by averaging the scores of the three items, summing these scores and dividing by 3. This method results in a score range from a minimum of 1 to a maximum of 4.
  units on a scale | 2.31 (.98) | 2.45 (.94) | 2.75 (.94) | 2.16 (.97) | 2.50 (.97)

OUTCOME MEASURES:

1. Primary Outcome: Mean Susceptibility to Vaping Score
Description: The 3-item Susceptibility to Vaping Scale assesses the extent to which adolescents are open to vaping, using a 1 to 4 response option scale. Here, 1 indicates the lowest susceptibility to vaping, and 4 represents the highest, with higher values indicating a greater susceptibility to vaping - essentially, a worse outcome. The overall scale score is determined by averaging the scores of the three items, summing these scores and dividing by 3. This method results in a score range from a minimum of 1 to a maximum of 4.
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 2.16 (1.04) | 2.21 (1.01) | 2.36 (1.07)

2. Secondary Outcome: Mean Attention Score
Description: The 1-item mean attention measure assesses the extent to which a participant reports that an advertisement captures their attention. Response options range from 1 to 5, with higher scores indicating stronger attention, which is considered a better outcome.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 4.49 (.79) | 4.49 (.77) | 4.10 (1.11)

3. Secondary Outcome: Mean Negative Affect Score
Description: The 3-item Negative Affect Scale assesses the extent to which an advertisement elicits negative emotions from the participant, such as fear or disgust. Response options range from 1 to 5. The overall scale score is calculated by averaging the scores of the three items, resulting in a minimum possible score of 1 and a maximum of 5. Higher scores indicate stronger negative emotions. In the context of this assessment, higher negative emotions are considered a more effective (better) outcome.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 3.42 (1.13) | 3.19 (1.19) | 2.68 (1.33)

4. Secondary Outcome: Mean Cognitive Elaboration Score
Description: The 3-item Mean Cognitive Elaboration Scale assesses the extent to which participants have thought about the addictiveness or harmfulness of vaping over the past 7 days. Response options range from 1 to 5. The overall scale score is calculated by averaging the three items, with scores ranging from a minimum of 1 to a maximum of 5. Higher scores indicate greater cognitive elaboration, suggesting a more effective engagement with the content (a better outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 3.59 (1.20) | 3.57 (1.21) | 3.43 (1.28)

5. Secondary Outcome: Mean Social Interactions Score
Description: The 3-item Mean Social Interactions Scale assesses the extent to which a participant has discussed the addictiveness or harmfulness of vaping with others in the past 7 days. Response options range from 1 (0 times) to 6 (11 or more times). The overall scale score is calculated by averaging the three items, resulting in a score range from a minimum of 1 to a maximum of 6. Higher scores indicate more frequent social interactions, which are considered a better outcome.
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 3.33 (1.39) | 3.20 (1.36) | 3.19 (1.45)

6. Secondary Outcome: Mean Vaping Health Harm Risk Beliefs Score
Description: The 3-item Vaping Health Harm Risk Beliefs Scale assesses the extent to which participants believe that vaping will lead to health harms. Response options range from 1 to 5. The overall scale score is calculated by averaging the three items, with possible scores ranging from a minimum of 1 to a maximum of 5. Higher scores indicate stronger beliefs in the health risks associated with vaping, which is considered a better outcome.
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 4.09 (1.08) | 4.09 (1.03) | 3.85 (1.18)

7. Secondary Outcome: Mean Vaping Addiction Risk Beliefs Score
Description: The 3-item Vaping Addiction Risk Beliefs Scale assesses the extent to which participants believe that vaping will lead to addiction. Response options range from 1 to 5. The overall scale score is calculated by averaging the three items, with a score range from 1 to 5. Higher scores indicate stronger beliefs in the risk of addiction due to vaping, which is considered a better outcome.
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 3.77 (1.18) | 3.78 (1.13) | 3.58 (1.28)

8. Secondary Outcome: Mean Vaping Attitudes Score
Description: The 3-item Vaping Attitudes Scale assesses a participant's attitude towards vaping (e.g., good/bad). Response options range from 1 to 5. The overall scale score is calculated by averaging the three items, with scores ranging from 1 to 5. Higher scores indicate a more positive attitude toward vaping, which is considered a less desirable outcome (i.e., worse outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 2.35 (1.29) | 2.37 (1.25) | 2.60 (1.33)

9. Secondary Outcome: Number of Days Participants Vape (E-cigarette Use)
Description: Participants will be asked to report the number of days they vaped over the past 21 days. We chose to retain the continuous measure of the number of days spent vaping rather than dichotomizing this outcome, due to the substantial variability observed in the number of days e-cigarettes were used. A higher value indicates more days that participants vaped, which is considered a less desirable outcome (i.e., worse outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
days | 1.86 (2.08) | 1.98 (2.19) | 2.14 (2.11)

10. Secondary Outcome: Mean Smoking Health Harm Risk Belief Score
Description: The 1-item Mean Smoking Health Harm Risk Belief Measure assesses the extent to which a participant believes that smoking will lead to health harms. Response options range from 1 to 5, with higher scores indicating stronger beliefs in the health risks associated with smoking, which is considered a desirable outcome (i.e., better outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 4.02 (1.22) | 3.98 (1.28) | 3.83 (1.29)

11. Secondary Outcome: Mean Smoking Addiction Risk Belief Score
Description: The 1-item mean smoking health harm risk belief measure assesses the extent to which a participant believes that smoking will lead to health harms. Response options are on a 1 to 5 scale, with higher scores representing a stronger health harm beliefs about smoking, which is a desirable outcome (i.e., better outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 3.79 (1.33) | 3.82 (1.33) | 3.76 (1.37)

12. Secondary Outcome: Mean Smoking Attitude Score
Description: The 1-item mean smoking attitude measure assesses a participant's attitude toward smoking (i.e., good/bad). Response options are on a 1 to 5 scale, with higher scores representing a more positive attitude toward smoking, which is considered as less desirable outcome (i.e., worse outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 2.13 (1.38) | 2.16 (1.42) | 2.35 (1.46)

13. Secondary Outcome: Mean Susceptibility to Smoking Cigarettes
Description: The 3-item Mean Susceptibility to Smoking Cigarettes Scale assesses a participant's susceptibility to smoking cigarettes. Response options range from 1 to 5. The overall scale score is calculated by averaging the three items, with possible scores ranging from 1 to 5. Higher scores indicate a stronger susceptibility to smoking, which is considered a less desirable outcome (i.e., worse outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 2.02 (1.02) | 2.05 (1.02) | 2.21 (1.05)

14. Secondary Outcome: Number of Days That Participants Who Smoke Cigarettes
Description: Participants will be asked to report the number of days they smoked cigarettes over the past 21 days. We chose to retain the continuous measure of the number of days smoking rather than dichotomizing this outcome, due to the substantial variability observed in the number of days cigarettes were used. A higher value indicates more days that participants smoked cigarettes, which is considered a less desirable outcome (i.e., worse outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
days | 1.61 (1.94) | 1.63 (2) | 1.8 (1.96)

15. Other Pre Specified Outcome: Mean Perceived Message Effectiveness Score (UNC Youth Scale)
Description: The 3-item UNC Youth Mean Perceived Message Effectiveness Scale assesses a participant's judgment of an advertisement's impact on their vaping beliefs and behaviors. Response options range from 1 to 5. The overall score is calculated by averaging the three items, with possible scores ranging from 1 to 5. Higher scores indicate that participants perceive the advertisements as more effective (i.e., better outcome).
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 4.18 (.82) | 4.14 (.86) | 3.32 (1.36)

16. Other Pre Specified Outcome: Mean Perceived Message Effectiveness Score (FDA Scale)
Description: The 6-item FDA Mean Perceived Message Effectiveness Scale evaluates a participant's overall impressions of an advertisement. Responses are provided on a scale from 1 to 5. The overall scale score is calculated by averaging these six items, resulting in a possible range of 1 to 5. Higher scores indicate that participants found the advertisements to be more informative (i.e., better outcome).
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 4.38 (.63) | 4.35 (.63) | 4.10 (.86)

17. Other Pre Specified Outcome: Mean Avoidance Score
Description: The 3-item Avoidance Scale measures the degree to which a participant wishes to avoid engaging with an advertisement. Responses are provided on a scale from 1 to 5. The overall score is calculated by summing the scores of the three items and then dividing by 3, resulting in a possible range of 1 to 5. Higher scores indicate greater avoidance, which is considered a less desirable outcome (i.e., worse outcome).
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 2.74 (1.31) | 2.57 (1.30) | 2.58 (1.30)

18. Other Pre Specified Outcome: Mean Reactance Score
Description: The 1-item reactance measure evaluates the degree to which an ad annoys participants, using a response scale from 1 to 5. Higher scores indicate greater reactance to the ad, representing a less favorable outcome.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 2.39 (1.53) | 2.28 (1.48) | 2.25 (1.46)

19. Other Pre Specified Outcome: Mean Vaping Social Enhancement Beliefs Score
Description: The 3-item Mean Vaping Social Enhancement Beliefs Scale measures participants' perceptions of the social benefits of vaping, such as fitting in better with friends. Responses are on a 1 to 5 scale, with overall scores calculated by averaging the three items. Scores range from 1 to 5, where higher scores indicate a stronger belief in the social benefits of vaping, a less desirable outcome (i.e., worse outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 2.84 (1.29) | 2.93 (1.30) | 3.09 (1.31)

20. Other Pre Specified Outcome: Mean Vaping Affect Regulation Beliefs Score
Description: The 3-item Mean Vaping Affect Regulation Beliefs Scale evaluates participants' beliefs about the experiential benefits of vaping, such as feeling good. Responses are recorded on a 1 to 5 scale. The overall score, which also ranges from 1 to 5, is calculated by averaging the three items. Higher scores indicate that participants expect more significant emotional or affective benefits from vaping, which is considered a less desirable outcome (i.e., worse outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 3.24 (1.28) | 3.28 (1.30) | 3.46 (1.27)

21. Other Pre Specified Outcome: Mean Vaping Injunctive Norms Score
Description: The 3-item Mean Vaping Injunctive Norms Scale measures participants' perceptions of others' approval or disapproval of their vaping behavior, using a response scale from 1 to 5. Overall scores, which range from 1 to 5, are calculated by averaging the three items. Higher scores indicate stronger perceived disapproval of vaping, which is considered a desirable outcome (i.e., better outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
score on a scale | 4.27 (.86) | 4.26 (.90) | 4.18 (.93)

22. Other Pre Specified Outcome: Mean Vaping Refusal Self-efficacy
Description: The 3-item Mean Vaping Refusal Self-Efficacy Scale measures a participant's confidence in their ability to refuse vaping in social situations, with response options ranging from 1 to 5. The overall score, also ranging from 1 to 5, is calculated by averaging the three items. Higher scores indicate stronger self-efficacy beliefs in refusing vaping, which is considered a desirable outcome (i.e., better outcome).
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads
Number analyzed (Participants) | 504 | 506 | 504
units on a scale | 3.50 (1.06) | 3.53 (1.02) | 3.51 (1.12)

ADVERSE EVENTS:
Time Frame: 3 months
Description: The protocol does not require Adverse Event Collections and/or All-Cause Mortality data.
Arm/Group | The Real Cost Vaping Prevention Ads - Health Effects Theme | The Real Cost Vaping Prevention Ads - Addiction Theme | Neutral Vaping Ads | Pilot Trial Group
All-Cause Mortality (participants affected / at risk) | 0/504 | 0/506 | 0/504 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/504 | 0/506 | 0/504 | 0/51
Other Adverse Events (participants affected / at risk) | 0/504 | 0/506 | 0/504 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT04836455/Prot_001.pdf
  • Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT04836455/SAP_000.pdf